CLINICAL TRIAL: NCT02252497
Title: Tranexamic Acid in Total Hip Arthroplasty: Single Preoperative Administration vs Perioperative Administration. A Randomized Control Trial.
Brief Title: Tranexamic Acid in Total Hip Arthroplasty.
Acronym: PORTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1308015; 2013-000791-15 (EudraCT Number)
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Hip Arthroplasty
Keywords: hip arthroplasty; Tranexamic acid; randomized control trial
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator): * 1g Intra Venous just before surgery
  * Then infusion of 1g of Exacyl over eight hours.
  Interventions: Drug: Active comparator : Tranexamic Acid (Exacyl)
- Physiologic serum (Placebo Comparator): * 1g Intra Venous, just before surgery
  * Then infusion of 1g of physiologic serum over eight hours.
  Interventions: Drug: Placebo comparator : physiologic serum

INTERVENTIONS:
Drug: Active comparator : Tranexamic Acid (Exacyl) — * 1g Exacyl Intra Venous, just before surgery
  * Then infusion of 1g of Exacyl over eight hours .
  Arms: Tranexamic acid
Drug: Placebo comparator : physiologic serum — * 1g Intra Venous just before surgery
  * Then infusion of 1g of physiologic serum over eight hours
  Arms: Physiologic serum

SUMMARY:
The purpose of this study is to compare a single preoperative dose of 1g of tranexamic acid (TXA) versus a preoperative dose of 1g of TXA followed by a continuous infusion of 1g over height hours on blood loss.

DETAILED DESCRIPTION:
The purpose of this study is to compare a single preoperative dose of 1g of tranexamic acid (TXA) versus a preoperative dose of 1g of TXA followed by a continuous infusion of 1g over eight hours on blood loss. The efficacy of TXA on blood loss is greatly influenced by the timing of its administration relative to surgery. In total hip arthroplasty, TXA should be started before surgery. However the optimal duration of TXA administration in hip arthroplasty is unknown. Numerous studies have shown that a single preoperative administration of TXA is effective. Yet indirect comparisons indicate a higher efficacy of TXA started before surgery and followed with a continuous infusion or repeated boluses. Our hypothesis is that a single preoperative administration of TXA is not sufficient to maintain therapeutic concentrations of TXA in the postoperative period. In addition a pharmacokinetic/pharmacodynamic study will be performed to identify the contribution of TXA plasma concentration as a predictor of blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring hip arthroplasty in first line, except recent hip fracture (less than 3 months)
* Consent of the patient or a family member or the support person.

Exclusion Criteria:

* Contraindication to tranexamic acid.
* Contraindication to apixaban.
* Pregnancy.
* Patient receiving a curative anticoagulating treatment in the preoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Calculated volume of blood losses in the peroperative period. | between the beginning of surgery and the fifth day
  It requires the sampling of haemoglobin at the beginning of surgery and in the fifth day.

SECONDARY OUTCOMES:
the patients' percentage that will receive the transfusion of at least one allogenic globular sediment | between D1 (day of surgery) and D5 (the fourth postoperative day)
  the patients' percentage that will receive the transfusion of at least one allogenic globular sediment in the peroperative period.
incidence of symptomatic thrombotic events and death | in 6 weeks
  combined criteria of venous events (deep venous thrombosis or pulmonary embolism), arterial events (acute coronary syndrome, stroke or peripheral arterial thrombosis) and death
tranexamic acid pharmacokinetic analyses | from the beginning of surgery up to 8 hours
  non linear mixt effect model

CONTACTS AND LOCATIONS:
Overall Officials: Paul ZUFFEREY, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France